CLINICAL TRIAL: NCT07060820
Title: Association Between Radial Artery Access Point and Radial Artery Spasm During Transradial Procedures
Brief Title: Association Between Radial Artery Access Point and Radial Artery Spasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Medicalpark Hastanesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMP-KAR-VA-01
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Radial Artery Spasm
Keywords: Transradial Access; Radial Artery Spasm; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0-20 mm Puncture Distance Group (Experimental): Radial artery puncture performed 0-20 mm proximal to the radial styloid process during transradial coronary angiography to evaluate its effect on the incidence of radial artery spasm (RAS).
  Interventions: Procedure: Radial Artery Puncture at 0-20 mm
- 21 mm Puncture Distance Group (Experimental): Radial artery puncture performed 21-40 mm proximal to the radial styloid process during transradial coronary angiography to evaluate its effect on the incidence of radial artery spasm (RAS).
  Interventions: Procedure: Radial Artery Puncture at >21 mm

INTERVENTIONS:
Procedure: Radial Artery Puncture at 0-20 mm — Radial artery puncture performed 0-20 mm proximal to the radial styloid process during transradial coronary angiography to evaluate its impact on the incidence of radial artery spasm (RAS).
  Arms: 0-20 mm Puncture Distance Group
Procedure: Radial Artery Puncture at >21 mm — Radial artery puncture performed at a distance greater than 21 mm proximal to the radial styloid process during transradial coronary angiography to evaluate its impact on the incidence of radial artery spasm (RAS).
  Arms: 21 mm Puncture Distance Group

SUMMARY:
This prospective clinical study aims to investigate whether the puncture site distance from the radial styloid process affects the incidence of radial artery spasm (RAS) during coronary angiography. Patients undergoing coronary angiography via radial access will be randomized into two groups based on the puncture site distance: 0-20 mm and >21 mm from the styloid process. The procedure will be performed by experienced interventional cardiologists using standard techniques and medications. The primary goal is to determine if a specific puncture site reduces the incidence of RAS, which is a common complication during transradial procedures. The study will also record procedural details and monitor for other complications to identify the optimal puncture site for reducing RAS and improving patient comfort.

DETAILED DESCRIPTION:
The transradial approach (TRA) is the standard vascular access route for diagnostic coronary angiography and percutaneous coronary interventions, in accordance with contemporary guidelines, due to lower bleeding risk, improved patient comfort, and facilitation of early mobilization compared with femoral access. Despite these advantages, radial artery spasm (RAS) remains a common and clinically relevant complication during transradial procedures, often associated with procedural difficulty, the need for access site crossover, and patient discomfort.

RAS is characterised by sudden, transient contraction of the radial artery during sheath insertion or catheter manipulation, which may result in difficulty in catheter advancement, and, in rare cases, procedural failure or catheter entrapment. Several clinical and procedural factors have been identified as being associated with the development of RAS, including female sex, smaller arterial diameter, use of larger sheaths, inadequate sedation, and limited operator experience. Currently radial access is recommended near the styloid process but there is limited data on the effects of different puncture distances from the styloid process on the development of RAS. We examined the impact of different radial artery puncture distances from the styloid process, on the development of radial artery spasm and access-site-related complications.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years and older. Patients scheduled for coronary angiography via transradial access. Patients with a palpable radial artery pulse. Patients with a normal Allen test.

Exclusion Criteria:

Abnormal Allen test results. Absence of palpable radial artery pulse. History of prior transradial coronary angiography with hemodynamic instability. Patients with severe comorbid conditions precluding safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Radial Artery Spasm during Transradial Coronary Angiography | During the procedure
  İnsidance of Radial Artery Spasm during Transradial Coronary Angiography

SECONDARY OUTCOMES:
Incidence of access site complications | Within 5 days post-procedure
  Number of patients experiencing access site complications including hematoma, bleeding, or occlusion within 5 days after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Vedat ASLAN, MD, Principal Investigator — Toros University
Locations (1):
- VM Medicalpark Mersin Hospital, Mersin, Mezitli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a single-center observational procedural study with limited resources for external data sharing and monitoring. Data can be shared upon reasonable request to the principal investigator in compliance with local regulations.